CLINICAL TRIAL: NCT04721951
Title: CO2-EVAR - An Innovative Approach to Automated Carbon Dioxide Angiography During Endovascular Abdominal Aortic Aneurysm Repair - (Proof of Concept Study)
Brief Title: An Innovative Approach to Automated Carbon Dioxide Angiography During Endovascular Abdominal Aortic Aneurysm Repair
Acronym: CO2-EVAR
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Andrea Vacirca, MD, University of Bologna
Other Study IDs: CO2-EVAR
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Endovascular Aortic Repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular Aortic Repair using Carbon Dioxide Angiography — Endovascular Aortic Repair using Carbon Dioxide Angiography

SUMMARY:
The study aims to perform Endovascular Aortic Repair procedures with CO2-Angiography using a standardized an operative Protocol

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Male, female
* Patients with indication for AAA
* Informed consent achievement

Exclusion Criteria:

* Severe COPD (Chronic Obstructive Pulmonary Disease)
* Known atrium- or ventricular septal defect with right-left-shunt
* Severe renal arteries atherosclerosis
* Ruptured AAA
* Current partecipation in other interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with AAA, undergoing EVAR
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Technical Success | 30 Days
  Technical success to assess the renal ostia and the hypogastric arteries (defined as 100% accuracy correlated to the iodinated contrast agent angiography or IVUS/FUSION techniques)

SECONDARY OUTCOMES:
Image Quality | 30 Days
  Image quality for guiding the procedure defined as good for stent-graft implantation or low not allowing stent-graft implantation
Endoleak Detection | 30 Days
  Type I-IV endoleak detection
CO2 Quantity | 30 Days
  Amount of CO2 at each deployment step (renal arteries, right/left hypogastric artery, final angiography)
Aneurysm Exclusion | 30 Days
  Aneurysm exclusion without type I or III endoleaks at the CT scan at discharge
Adverse Events | 30 Days
  Any adverse event within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, Prof, Principal Investigator — Department of experimental diagnostic and specialty medicine - Vascular Surgery - University of Bologna
Locations (1):
- Department of experimental diagnostic and specialty medicine - Vascular Surgery, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided